CLINICAL TRIAL: NCT00116935
Title: Short (12 Months) Versus Long (36 Months) Duration of Adjuvant Treatment With the Tyrosine Kinase Inhibitor Imatinib Mesylate of Operable GIST With a High Risk of Recurrence
Brief Title: Study Comparing 12 Months Versus 36 Months of Imatinib in the Treatment of Gastrointestinal Stromal Tumor (GIST)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Scandinavian Sarcoma Group (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SSGXVIII/AIO
Record Dates: First submitted 2005-06-30; First posted 2005-07-01 (Estimated); Last update posted 2011-12-30 (Estimated); Status verified 2011-12

CONDITIONS: Sarcoma
Keywords: Gastrointestinal stromal tumor; GIST; Sarcoma; Imatinib; Adjuvant therapy; KIT; PDGFRA; Receptor tyrosine kinase; Tyrosine kinase inhibitor
MeSH Terms: conditions — Sarcoma; Gastrointestinal Stromal Tumors | interventions — Imatinib Mesylate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): 1 year of adjuvant imatinib mesylate 400 mg/day orally
  Interventions: Drug: imatinib mesylate; Drug: imatinib
- 2 (Experimental): 3 years of adjuvant imatinib mesylate 400 mg/day orally
  Interventions: Drug: imatinib

INTERVENTIONS:
Drug: imatinib mesylate — imatinib 400 mg/day orally qd for 12 months
  Other Names: Gleevec
  Arms: 1
Drug: imatinib — imatinib 400 mg/d orally qd for 36 months
  Other Names: Gleevec
  Arms: 1
Drug: imatinib — imatinib 400 mg/d orally qd for 36 months
  Other Names: Gleevec
  Arms: 2

SUMMARY:
In this study, patients who have been diagnosed with gastrointestinal stromal tumor (GIST) will be randomly allocated in a 1:1 ratio to receive imatinib (Gleevec) either for 12 or for 36 months following surgery. The study participants are required to have a histologically verified GIST with a high risk of GIST recurrence despite complete removal of all macroscopic GIST tissue at surgery. The high/very high risk of recurrence is defined as one of the following: 1) the largest tumor diameter is over 10 cm; 2) the mitosis count is high (over 10 mitoses per 50 high power microscope fields, HPFs); 3) the largest tumor diameter over 5 cm and the mitosis count is over 5/50 HPFs; 4) tumor spillage has taken place into the abdominal cavity at the time of surgery or following spontaneous tumor rupture. All study participants will receive imatinib 400 mg/day orally, but the duration of imatinib administration will be determined randomly (either for 12 or for 36 months). The study participants will be followed up using blood tests and computed tomography (or MRI) of the abdomen. The computed tomography examinations will be performed at 6 month intervals for a median of 5 years. A total of 280 patients will be entered into the study. The study hypothesis is that adjuvant imatinib may prevent some of the GIST recurrences, and that there may be a difference in the rate of GIST recurrence between the two groups.

DETAILED DESCRIPTION:
This is an open-label, randomized, prospective, phase III, multicenter study carried out in the Nordic countries and in Germany. Following macroscopically complete surgery, the study participants will be allocated to receive imatinib either for 12 or for 36 months. At randomization, the patients are stratified into 2 strata: 1) local disease (1 GIST tumor); 2) intra-abdominal implants or resectable intra-abdominal/hepatic metastases, or intra-abdominal spillage is present, or R1 surgery has been carried out (microscopic disease has been left behind). The imatinib dose is 400 mg/day administered with food. Imatinib dose adjustments are made as per protocol.

Medical history, current medication, weight, height, and ECOG performance status are recorded prior to study entry. Physical examination, blood cell counts, blood biochemistry, pregnancy test, chest X-ray or CT, and CT or MRI of the abdomen and pelvis are carried out/measured prior to study entry. FDG-PET is an optional staging examination. Research serum samples are collected for banking prior to initiating imatinib and at 6-month intervals during the study. Tumor tissue is reviewed centrally to confirm the histological diagnosis of GIST, and KIT and PDGFRA gene mutation analyses will be performed from stored GIST tissue.

The study participants are monitored during adjuvant treatment and following adjuvant treatment. Physical examination, weight and ECOG performance status are assessed at 4- to 26-week intervals. Adverse events are collected using structured forms at the times of the evaluation visits. Blood cell counts and blood biochemistry are measured at 2- to 6-week intervals during imatinib therapy, and at 6-month intervals following completion of adjuvant therapy. CT or MRI examinations of the abdomen and pelvis are performed at 6-month intervals during the study.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* Histologically documented diagnosis of GIST
* Resectable GIST
* GIST removed at open surgery
* Immunohistochemical documentation of GIST (immunostaining for KIT/CD117)
* High risk of tumor recurrence as defined as one of the following: 1) the largest tumor diameter greater than 10.0 cm (measured by a pathologist, with any mitotic count); 2) mitotic count over 10 mitoses per 50 high power fields (HPFs) (with any tumor size); the largest tumor diameter larger than 5.0 cm and the mitotic count is over 5/50 HPFs; 4) tumor spillage into the abdominal cavity at surgery (or tumor rupture). No residual tumors must be present at laparotomy, or in postoperative CT or MRI examinations. Patients who have microscopically infiltrated margins (or suspected microscopical infiltration, R1) are also allowed to enter study.
* Performance status 0, 1, or 2 (ECOG)
* Adequate organ function, defined as follows: total bilirubin <1.5 x ULN (upper limit of normal), serum AST (SGOT) and ALT (SGPT) <2.5 x ULN, creatinine <1.5 x ULN, ANC (neutrophil count) >1.5 x 10^9/L, platelets >100 x 10^9/L.
* Negative pregnancy test (females with childbearing potential)
* Written, voluntary informed consent

Exclusion Criteria:

* Inoperable or metastatic GIST
* Less than 1 week or more than 12 weeks has elapsed from surgery
* Recurrent GIST
* Patient has received any investigational agents within 28 days as calculated from the first day of the study drug dosing
* Patient is less than 5 years free from another primary malignancy
* Patient with grade III/IV cardiac problems as defined by the New York Heart Association Criteria
* Female patients who are pregnant or breast-feeding
* Patient has severe or uncontrolled medical disease (i.e. uncontrolled diabetes, severe chronic renal disease, or active uncontrolled infection). Concurrent use of warfarin or acetaminophen are not allowed with imatinib.
* Chronic liver disease
* Known diagnosis of human immunodeficiency virus (HIV) infection
* Patient has received chemotherapy for GIST
* Patient has received neoadjuvant imatinib therapy prior to randomization
* Radiotherapy to 25% or more of the bone marrow
* Patient with any significant history of non-compliance to medical regimens or with inability to grant reliable informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2004-02; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Recurrence-free survival | 5 years

SECONDARY OUTCOMES:
Adverse effects | 5 years
Survival | 5 years
GIST-specific survival | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Heikki Joensuu, M.D., Principal Investigator — Department of Oncology, Helsinki University Central Hospital
Locations (1):
- Scandinavian Sarcoma Group, Southern Swedish Regional Tumour Registry, Lund University Hospital, Lund, Sweden

REFERENCES:
- [Derived] Joensuu H, Reichardt A, Eriksson M, Hohenberger P, Boye K, Cameron S, Lindner LH, Jost PJ, Bauer S, Schutte J, Lindskog S, Kallio R, Jaakkola PM, Goplen D, Wardelmann E, Reichardt P. Survival of patients with ruptured gastrointestinal stromal tumour treated with adjuvant imatinib in a randomised trial. Br J Cancer. 2024 Jul;131(2):299-304. doi: 10.1038/s41416-024-02738-z. Epub 2024 Jun 11. PMID 38862742
- [Derived] Joensuu H, Eriksson M, Sundby Hall K, Reichardt A, Hermes B, Schutte J, Cameron S, Hohenberger P, Jost PJ, Al-Batran SE, Lindner LH, Bauer S, Wardelmann E, Nilsson B, Kallio R, Jaakkola P, Junnila J, Alvegard T, Reichardt P. Survival Outcomes Associated With 3 Years vs 1 Year of Adjuvant Imatinib for Patients With High-Risk Gastrointestinal Stromal Tumors: An Analysis of a Randomized Clinical Trial After 10-Year Follow-up. JAMA Oncol. 2020 Aug 1;6(8):1241-1246. doi: 10.1001/jamaoncol.2020.2091. PMID 32469385
- [Derived] Joensuu H, Wardelmann E, Sihto H, Eriksson M, Sundby Hall K, Reichardt A, Hartmann JT, Pink D, Cameron S, Hohenberger P, Al-Batran SE, Schlemmer M, Bauer S, Nilsson B, Kallio R, Junnila J, Vehtari A, Reichardt P. Effect of KIT and PDGFRA Mutations on Survival in Patients With Gastrointestinal Stromal Tumors Treated With Adjuvant Imatinib: An Exploratory Analysis of a Randomized Clinical Trial. JAMA Oncol. 2017 May 1;3(5):602-609. doi: 10.1001/jamaoncol.2016.5751. PMID 28334365
- [Derived] Joensuu H, Eriksson M, Sundby Hall K, Reichardt A, Hartmann JT, Pink D, Ramadori G, Hohenberger P, Al-Batran SE, Schlemmer M, Bauer S, Wardelmann E, Nilsson B, Sihto H, Bono P, Kallio R, Junnila J, Alvegard T, Reichardt P. Adjuvant Imatinib for High-Risk GI Stromal Tumor: Analysis of a Randomized Trial. J Clin Oncol. 2016 Jan 20;34(3):244-50. doi: 10.1200/JCO.2015.62.9170. Epub 2015 Nov 2. PMID 26527782
- [Derived] Joensuu H, Eriksson M, Sundby Hall K, Hartmann JT, Pink D, Schutte J, Ramadori G, Hohenberger P, Duyster J, Al-Batran SE, Schlemmer M, Bauer S, Wardelmann E, Sarlomo-Rikala M, Nilsson B, Sihto H, Monge OR, Bono P, Kallio R, Vehtari A, Leinonen M, Alvegard T, Reichardt P. One vs three years of adjuvant imatinib for operable gastrointestinal stromal tumor: a randomized trial. JAMA. 2012 Mar 28;307(12):1265-72. doi: 10.1001/jama.2012.347. PMID 22453568
- See also: Scandinavian Sarcoma Group web site — http://www.ssg-org.net